CLINICAL TRIAL: NCT00821158
Title: The DIEP Flap as a Model of Ischemia-Reperfusion: an Intervention Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: R. van der Hulst, M.D., Phd, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEC 25-11-2008
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Ischemia-Reperfusion
MeSH Terms: interventions — Antioxidants; Anti-Inflammatory Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo tablet and iv
  Interventions: Other: Placebo
- 2 (Experimental): Placebo tablet and intervention iv
  Interventions: Drug: Antioxidant
- 3 (Experimental): Intervention tablet and placebo iv
  Interventions: Drug: Anti-inflammatory drug

INTERVENTIONS:
Drug: Antioxidant — Antioxidant iv bolus
  Arms: 2
Other: Placebo — Placebo tablet and iv
  Arms: 1
Drug: Anti-inflammatory drug — Anti-inflammatory tablet
  Arms: 3

SUMMARY:
The investigators will examine whether administration of certain medications will decrease or prevent ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing breast reconstruction

Exclusion Criteria:

* Diabetes mellitus
* Kidney or liver disease
* Use of immunosuppressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Antioxidant concentrations | 0,5-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: R. van der Hulst, M.D., Phd, Study Chair — Maastricht Universtity Medical Center; Marieke van den Heuvel, M.D., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands